CLINICAL TRIAL: NCT03468309
Title: Medication Optimization Using Pharmacogenetic Testing and the Genomind Drug Interaction Guide (G-DIG) to Reduce Polypharmacy in a Mental Health Population
Brief Title: Medication Optimization Using Pharmacogenetic Testing and the G-DIG to Reduce Polypharmacy in a Mental Health Population
Acronym: MedOPT
Status: Completed | Type: Observational
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Genomind, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 01600
Record Dates: First submitted 2017-11-16; First posted 2018-03-16 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-02

CONDITIONS: Pharmacogenetic Testing
Keywords: polypharmacy; drug interactions; DNA testing; mental health diagnosis; drug side effects; presciption treatment plans; mental health medication treatment plans
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a cheek swab tissue sample for DNA collection will be obtained from each consented study participant in order to complete the pharmacogenomic testing; via the Genecept Assay testing results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genecept Assay and G-DIG decision tool: Veterans who have been prescribed 5 or more medications, with at least two being for a mental health diagnosis. Also allowable would be one medication for a mental health diagnosis and another medication for side effects related to a medication prescribed for the mental health diagnosis.
  Interventions: Genetic: Genecept Assay and G-DIG decision tool

INTERVENTIONS:
Genetic: Genecept Assay and G-DIG decision tool — Participating providers will review results of the Genecept Assay using a secure web-based program and will utilize the G-DIG tool in order to determine the optimal medication regime for the patient, based on their individual genetic profile. Genomind will provide training to all investigators prior to the study start regarding the interpretation of the pharmacological assay and the use of the G-DIG tool. Genomind representatives will be available throughout the duration of the study for consultation regarding the interpretation and implementation of the testing results. All final decisions about changing dosage, adding medications, or removing medications will be determined by the provider.

SUMMARY:
Use of polypharmacy has significantly increased over the past two decades, which has unproven clinical benefit and is associate with an increased the risk of adverse side effects. Pharmacogenetic assays, such as the Genecept® Assay, have the purported benefit of being able to predict response(s) to specific medication based on genetic markers. Thus, this study is a 12-week open-label, naturalistic study of the provision of pharmacogenetic testing and a computerized decision tool for providers to determine the potential efficacy of the assay to reduce polypharmacy and improve patient outcomes.

DETAILED DESCRIPTION:
Use of polypharmacy has significantly increased over the past two decades, which has unproven clinical benefit and increased the risk of drug-drug interactions and adverse side effects. Pharmacogenetic assays have the purported benefit of being able to predict response(s) to specific medication based on genetic markers. One such assay is the Genecept® Assay produced by Genomind, which detects 63 allele polymorphisms of 18 genes. In addition, Genomind has developed the Genomind Drug Interaction Guide (G-DIG), which examines drug-drug-gene interactions. This computerized decision tool for medication providers uses the genetic information from the Genecept® Assay to look at the current medications being utilized to determine if there are specific drug-drug interactions that may be relevant given the individual's specific genetic test results.

This is a 12-week open-label, naturalistic study of the provision of pharmacogenetic testing information to both providers and patients. Fifty Veterans within the VAPSHCS who are prescribed polypharmacy, as defined as five or more medications, with at least two prescribed for a mental health diagnosis, and have a sub-optimal treatment effect will be enrolled in this study. Participating subjects will sign informed consent and a sample will be obtained in order to complete the pharmacogenomic testing. Medication providers who are participating in this study will utilize the pharmacogenetic assay results along with the G-DIG tool to design an optimized medication regime. The overall global level of symptoms and other patient symptoms measures will be administered at baseline, 6-weeks, and 12-weeks. The provider's medication plans will be compared before and after the pharmacogenetic assay information is provided. Number of medications will be reviewed to determine any reduction in polypharmacy and healthcare costs. The clinical global improvement scale (CGI) and patient assessments, including measures of depression, anxiety, PTSD, insomnia, pain, drug and alcohol use, quality of life, side effects, and medication adherence will be administered at baseline, 6-weeks, and 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Currently receiving outpatient care for mental health diagnosis at VA Puget Sound Health Care System (VA PSHCS) and referred by sub-investigator on listed for study
2. Currently experiencing a sub-optimal medication response as assessed by either continue symptoms or medication side effects; which in the opinion of their treating provider would indicate or warrant a change in medications
3. Currently prescribed at least five medications; two being for a mental health diagnosis OR one mental health medication prescribed for mental health diagnosis and one for mediating side effects related to the medication prescribed for the mental health diagnosis.
4. Between the ages of 18-75.

Exclusion Criteria:

1. Any mental health or physical health diagnosis, which in the opinion of their treating prescriber would prevent them from being compliant on a medication regimen or being able to complete the study measures.
2. Current/active diagnosis of severe alcohol or drug use disorder
3. Serious medical or mental health symptoms requiring immediate stabilization and/or hospitalization
4. Impaired decision making capacity that in the clinical judgment of their provider would affect their ability to provide informed consent
5. Self-identification as being current pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject pool will be drawn from Veterans receiving care at VA Puget Sound Health Care System for mental health diagnosis between the ages of 18-75 who meet all of the inclusion criteria with no indicators to any of the exclusionary criteria.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Wood, PhD., Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wood AE, Agrawal D, Deem AP, Dupper Knoper TL, Merino RF, Molzof HE, Maus LE, Kim F, Lodin Z, Lim S. Medication Optimization Using Pharmacogenomic Testing in a Complex Mental Health Population Prescribed Psychiatric Polypharmacy. J Clin Pharmacol. 2022 Jul;62(7):898-904. doi: 10.1002/jcph.2032. Epub 2022 Mar 4. PMID 35075665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment lasted from 10/04/2017 to 12/31/2018
Groups:
- Genecept Assay and G-DIG Decision Tool: Veterans prescribed 5 or more medications, with at least two being for a mental health diagnosis. Also allowable would be one medication for a mental health diagnosis and another for side effects related to a medication prescribed for the mental health diagnosis.
  Genecept Assay and G-DIG decision tool: Participating providers review results of the Genecept Assay using a secure web-based program and utilize the G-DIG tool to determine the optimal medication regime for the patient, based on their individual genetic profile. Genomind will provide training to all investigators prior to the study start regarding the interpretation of the pharmacological assay and the use of the G-DIG tool. Genomind representatives will be available throughout the duration of the study for consultation regarding the interpretation and implementation of the testing results. All final decisions about changing dosage, adding medications, or removing medications will be determined by the provider.
Period: Overall Study
Arm/Group | Genecept Assay and G-DIG Decision Tool
Started | 53
Completed | 47
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Participants as described in data tables.
Groups:
- Genecept Assay and G-DIG Decision Tool: Veterans prescribed 5 or more medications, with at least two being for a mental health diagnosis. Also allowable would be one medication for a mental health diagnosis and another for side effects related to a medication prescribed for the mental health diagnosis.
  Genecept Assay and G-DIG decision tool: Participating providers review results of the Genecept Assay using a secure web-based program and utilize the G-DIG tool to determine the optimal medication regime for the patient, based on their individual genetic profile. Genomind will provide training to all investigators prior to the study start regarding the interpretation of the pharmacological assay and the use of the G-DIG tool. Genomind representatives will be available throughout the duration of the study for consultation regarding the interpretation and implementation of the testing results. All final decisions about changing dosage, adding or removing medications will be determined by the provider.
Arm/Group | Genecept Assay and G-DIG Decision Tool
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 36
  More than one race | 7
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53
CGI [Mean (Standard Deviation); unit: units on a scale] | 4.07 (.62)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression
Description: Clinical Global Impression. Range is 1-6, with 1 = less symptomology and 6 = high symptomology.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genecept Assay and G-DIG Decision Tool
Number analyzed (Participants) | 50
units on a scale
  CGI at baseline | 4.07 (.62)
  CGI at 12-weeks | 3.96 (.59)
Statistical Analysis 1: Comparison: Genecept Assay and G-DIG Decision Tool; Test type: Superiority — T-test was used to compare means at baseline and 12-weeks; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Number of Psychiatric Medications
Description: Number of psychiatric medications prescribed to the patient.
Time Frame: Change from baseline to 12-weeks
Measure: Mean (Standard Deviation); unit: prescriptions
Arm/Group | Genecept Assay and G-DIG Decision Tool
Number analyzed (Participants) | 50
prescriptions
  Psychiatric meds at baseline | 3.85 (1.41)
  Psychiatric meds at 12-weeks | 3.70 (1.37)
Statistical Analysis 1: Comparison: Genecept Assay and G-DIG Decision Tool; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Patient Health Questionnaire-9 is a scale of depression, scores range from 0-27, with 0 representing less depression and 27 representing more depression.
Time Frame: Change from baseline to 12-weeks
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Genecept Assay and G-DIG Decision Tool
Number analyzed (Participants) | 50
scores
  PHQ-9 at baseline | 15.81 (5.68)
  PHQ-9 at 12-weeks | 13.43 (6.39)
Statistical Analysis 1: Comparison: Genecept Assay and G-DIG Decision Tool; Test type: Superiority; p < 0.05, ANOVA; Assumption of sphericity had been violated X2(2)=13.61, p<.01 so Huynh-Feldt correction was used

4. Secondary Outcome: Generalized Anxiety Scale-7 (GAD-7)
Description: Generalized Anxiety Scale-7 is a measure of anxiety, scores range from 0-21, with 0 representing less anxiety and 7 representing more anxiety.
Time Frame: Change from baseline to 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genecept Assay and G-DIG Decision Tool
Number analyzed (Participants) | 50
units on a scale
  GAD-7 at baseline | 13.60 (5.53)
  GAD-7 at 12-weeks | 12.02 (5.90)
Statistical Analysis 1: Comparison: Genecept Assay and G-DIG Decision Tool; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Baseline, 6-weeks, 12-weeks
Description: This is a naturalistic study, side effects of medication treatment are an expected part of treatment as usual and will be handled by their provider as part of their regular clinical care. A brief measure of side effects will be collected by patient interview at baseline, 6-weeks, and 12-weeks. If the participant reveals an emergent mental or physical health issue they will be treated as per clinical guidelines at the VA.
Arm/Group | Genecept Assay and G-DIG Decision Tool
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03468309/Prot_SAP_000.pdf